CLINICAL TRIAL: NCT07147868
Title: Effect of Education for Relatives of Chemotherapy Patients on Family Health, Nutrition, and Psychological Well-Being
Brief Title: Education for Chemotherapy Patients' Kin: Effects on Family Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Muhammet Faruk Yigit, Assistant Prof. Dr., Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10.02.2025-182158
Record Dates: First submitted 2025-08-15; First posted 2025-08-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Caregiver Awareness; Family Health; Psychological Well-being; Chemotherapy
Keywords: Chemotherapy; caregiver education; family health; psychological well-being; nutrition
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to intervention or control groups and assessed at baseline, mid-intervention, and post-intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Structured Caregiver Education Arm 2 (Control): No Structured Education (Experimental): Arm Type: Experimental Relatives of chemotherapy patients received a structured training program covering self-efficacy, nutrition, and stress management. The training was delivered in group sessions supported by educational materials.
  Interventions: Behavioral: Structured Education Program for Caregivers of Chemotherapy Patients
- Control Group (No Intervention) (No Intervention): Relatives of chemotherapy patients received standard care without additional structured training.

INTERVENTIONS:
Behavioral: Structured Education Program for Caregivers of Chemotherapy Patients — A structured educational intervention designed for caregivers of cancer patients undergoing chemotherapy, delivered in 30-45 minute sessions to groups of 4-5 participants. The program includes modules on self-efficacy, stress management, healthy lifestyle behaviors, interpersonal relationships, and nutrition based on the Mediterranean diet. Content covers evidence-based strategies for improving family health, psychological well-being, and dietary adherence. Sessions are conducted by a certified practitioner with 480 hours of family counseling training in a university hospital's medical oncology unit seminar room. The intervention aims to reduce caregiver burden, enhance psychological well-being, improve adherence to the Mediterranean diet, and promote family health, as assessed by the Family Health Scale (ASÖ), Mediterranean Diet Adherence Scale (MEDAS), and Psychological Well-Being Scale (PİO) at baseline (t0), post-intervention (t1), and 6 weeks follow-up (t2).
  Arms: Arm 1 (Experimental): Structured Caregiver Education Arm 2 (Control): No Structured Education

SUMMARY:
Aim: To evaluate the effects of structured education provided to the relatives of chemotherapy patients on family health, nutrition, and psychological well-being.

Methods: This randomized controlled study will be conducted with a parallel-group, pretest-posttest design at a university hospital in the northeastern region of Turkey. A total of 68 patient relatives are planned to participate (Intervention: 34, Control: 34). The training to be provided to the intervention group will cover topics such as self-efficacy, nutrition, and stress management. Data will be collected at three different time points (pretest, mid-test, posttest) using the Family Health Scale (FHS), the Mediterranean Diet Adherence Screener (MEDAS), and the Psychological Well-Being Scale (PWB). Statistical analyses will include chi-square tests, t-tests, and Pearson correlation coefficients.

DETAILED DESCRIPTION:
Aim: This study will evaluate the effects of structured education provided to the relatives of patients undergoing chemotherapy on family health, nutritional habits, and levels of psychological well-being.

Methods: The study is designed as a randomized controlled trial with a parallel-group, pretest-posttest design. It is planned to be conducted at a university hospital located in the northeastern region of Turkey, with a total of 68 patient relatives participating (Intervention Group: n = 34, Control Group: n = 34). The training materials will be developed to cover topics such as self-efficacy, nutrition, and stress management. Data will be collected using a participant information form, the Family Health Scale (FHS), the Mediterranean Diet Adherence Screener (MEDAS), and the Psychological Well-Being Scale (PWB) at three time points: t0 (pretest), t1 (mid-test), and t2 (posttest). Statistical analyses will include chi-square tests, paired sample t-tests for repeated measures, and Pearson correlation coefficients.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver (first-degree relative or emotional supporter) of a patient receiving chemotherapy.
* Age 18 years or older.
* Ability to read and understand Turkish.
* Provides care or emotional support to the chemotherapy patient.
* No chronic health conditions.
* Not receiving psychiatric treatment.
* No substance use.

Exclusion Criteria:

* Presence of cognitive or sensory impairments.
* Failure to attend at least two education sessions (for intervention group).
* Pregnancy.
* Voluntary withdrawal from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Psychological Well-Being Score | Baseline (t0), immediately post-intervention (t1), and 6 weeks post-intervention (t2).
  Description: Change in psychological well-being of caregivers, measured using the Psychological Well-Being Scale, an 8-item, 7-point Likert scale (scores range from 8 to 56, higher scores indicate better well-being). The scale assesses life satisfaction, stress coping, and positive emotions.
Mediterranean Diet Adherence Score | Time Frame: Baseline (t0), immediately post-intervention (t1), and 6 weeks post-intervention (t2).
  Change in adherence to the Mediterranean diet among caregivers, measured using the Mediterranean Diet Adherence Scale, a 14-item scale (scores range from 0 to 14, higher scores indicate greater adherence). Scores ≥7 indicate acceptable adherence, and ≥9 indicate high adherence.
Family Health Score | Baseline (t0), immediately post-intervention (t1), and 6 weeks post-intervention (t2).
  Change in family health levels among caregivers, measured using the Family Health Scale (FHS), short form (FHS-SF), a 10-item scale (scores range from 10 to 50, dichotomized to 0-10 for evaluation: 0-5 = poor, 6-8 = moderate, 9-10 = excellent family health).

SECONDARY OUTCOMES:
Correlation Between Psychological Well-Being and Family Health | Baseline (t0), immediately post-intervention (t1), and 6 weeks post-intervention (t2).
  Assessment of the relationship between psychological well-being and family health among caregivers, measured using Pearson correlation analysis to evaluate the strength and direction of the association.
Correlation Between Psychological Well-Being and Mediterranean Diet Adherence | Baseline (t0), immediately post-intervention (t1), and 6 weeks post-intervention (t2).
  Assessment of the relationship between psychological well-being and Mediterranean diet adherence among caregivers, measured using Pearson correlation analysis to evaluate the strength and direction of the association.
Correlation Between Family Health and Mediterranean Diet Adherence | Baseline (t0), immediately post-intervention (t1), and 6 weeks post-intervention (t2).
  Assessment of the relationship between family health and Mediterranean diet adherence among caregivers, measured using Pearson correlation analysis to evaluate the strength and direction of the association.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University Hospital, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers. The study collected sensitive data, including sociodemographic information, psychological well-being scores, Mediterranean diet adherence scores, and family health scores, from caregivers of chemotherapy patients. Data sharing is not planned due to privacy and ethical considerations, as participant confidentiality is protected under the ethical approvals obtained from the X University Health Sciences Research and Publication Ethics Committee and in accordance with the Helsinki Declaration.

REFERENCES:
- [Result] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- See also: link address — https://pubmed.ncbi.nlm.nih.gov/38572751/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT07147868/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT07147868/ICF_001.pdf